CLINICAL TRIAL: NCT06886607
Title: The Effects of Mindfulness and Web-Based Physical Activity Program on Mental and Cardiovascular Risk in Patients With Schizophrenia: A Randomized Controlled Trial
Brief Title: The Effects of Mindfulness and Web-Based Physical Activity Program in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Neslihan Lok, Prof.Dr, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SelcukU-GUzun-001
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia Disorders
Keywords: Schizophrenia; Mindfulness and web-based physical activity program; mental well-being; sleep quality; coping with stress; cardiovascular risk
MeSH Terms: conditions — Schizophrenia; Psychological Well-Being; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study was a randomized controlled trial with pre-test and post-test control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group was a group of 25 people consisting of patients with schizophrenia who followed the 14-week Mindfulness and Web-Based Physical Activity Program.
  Interventions: Behavioral: the Mindfulness and Web-Based Physical Activity Program
- Control (No Intervention): No intervention was applied to the control group throughout the 14-week program; the patients continued with their daily routine activities.

INTERVENTIONS:
Behavioral: the Mindfulness and Web-Based Physical Activity Program — The "Mindfulness and Web-Based Physical Activity Program" consists of two phases: the "Mindfulness Skill Development Program" and the "Mindful Physical Activity Program". In the first phase of the Program, the "Mindfulness Skill Development Program" was implemented for two weeks, five days a week, from October 23 to November 3, 2023. The program includes activities for individuals to develop mindfulness skills through videos uploaded on the YouTube channel. In the second phase of the Program, The 12-week Mindful Physical Activity Program, implemented between November 2023 and January 2024, consisted of "Mindful Walking" and "Mindful Physical Activity Day" sessions held twice a week (Tuesday and Thursday) and three days a week for 50 minutes. Each session began with a 10-minute warm-up exercise, followed by 40 minutes of endurance and strength training sessions, and ended with 10 minutes of cool-down exercises.
  Arms: Intervention

SUMMARY:
This study was aimed to examine the effects of the Mindfulness and Web-Based Physical Activity Program - consisting of two weeks of mindfulness skills followed by 12 weeks of walking and exercise - delivered through videos uploaded to a YouTube channel on mental and cardiovascular risk in patients with schizophrenia. The main questions it aims to answer are:

After the Mindfulness and Web-Based Physical Activity Program, H1-1: There is a statistically significant difference in the mean total scores of mental well-being between the intervention and control groups.

H1-2: There is a statistically significant difference in the mean total scores of sleep quality between the intervention and control groups.

H1-3: There is a statistically significant difference in the mean total scores of the subscales of the Coping Style Scale (self-confident approach, optimistic approach, helpless approach, submissive approach, and seeking of social support) between the intervention and control groups.

H1-4: There is a statistically significant difference in terms of cardiovascular risk levels between the intervention and control groups.

Researchers were compared the Mindfulness and Web-Based Physical Activity Program to a control group (no intervention) to see if the Mindfulness and Web-Based Physical Activity Program works on mental and cardiovascular risk in patients with schizophrenia.

Participants were:

* followed in the first phase of the Mindfulness and Web-Based Physical Activity Program, the "Mindfulness Skill Development Program", which included activities for individuals to develop their mindfulness skills, five days a week for two weeks from October 23 to November 3, 2023 through videos uploaded on the YouTube channel.
* followed in the second phase of the Mindfulness and Web-Based Physical Activity Program, the 12-week "Mindful Physical Activity Program", which consisted of "Mindful Walking" and "Mindful Physical Activity Day" sessions held twice a week (Tuesday and Thursday) and three days a week for 50 minutes from November 2023 to January 2024 through videos uploaded on the YouTube channel.

DETAILED DESCRIPTION:
The study included 110 individuals aged 25-55 who were diagnosed with schizophrenia and applied to the S.U. Faculty of Medicine Mental Health and Diseases Polyclinic in the last year, and were examined according to the inclusion-exclusion criteria. A total of 50 individuals were included in the study. These individuals were randomly assigned to two groups: intervention and control. Pre-test data were collected using the "Personal Information Form", "Mental Well-Being Scale", "Pittsburgh Sleep Quality Index (PSQI)", "Coping Style Scale", and "QRISK3 Index" from the intervention and control groups by researchers between October 2023 and January 2024 in the Group Therapy Room of the Mental Health and Diseases Polyclinic, based on self-reporting. The "Mindfulness and Web-Based Physical Activity Program" was completed in a total of 14 weeks, consisting of a 2-week "Mindfulness Skill Development Program" and a 12-week "Mindful Physical Activity Program" to intervention group through videos uploaded on the YouTube channel opened via the web. Before starting the Mindful Physical Activity Program, all participants in the intervention group were provided with sports shoes, resistance bands, exercise mats, and pedometers to encourage regular participation in physical activity. Additionally, the researchers gave participants the Mindful Physical Activity Program Follow-up Form and the Mindful Walking Follow-up Form to track their daily involvement in the program. At the end of the Mindfulness and Web-Based Physical Activity Program, both the intervention and control groups were administered the "Mental Well-Being Scale", "Pittsburgh Sleep Quality Index-PSQI", "Coping Style Scale", and "QRISK3 Index". No intervention was applied to the control group throughout the 14-week program; the patients continued with their daily routine activities.

ELIGIBILITY:
Inclusion Criteria:

* Being registered at the Mental Health and Illnesses Outpatient Clinic of S.U. Faculty of Medicine Hospital,
* Having been diagnosed with schizophrenia for at least 1 year
* Being between the ages of 25 and 55,
* Having scored mild to moderate on the Positive and Negative Syndrome Scale (PANSS)
* Having access to technological devices such as smartphones, computers, and tablets to watch videos from a YouTube channel.

Exclusion Criteria:

* Having physical, mental, visual, or hearing disabilities,
* Being involved in a program similar to the intervention to be applied,
* Having a condition that would prevent them from exercising,
* Having a diagnosis of heart disease or stroke.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Mental Well-Being total mean score | From enrollment to the end of the Mindfulness and Web-Based Physical Activity Program at 14 weeks
  The Mental Well-Being Scale scores range from 14 to 70 points. A higher score on the scale indicates a higher level of mental well-being.
Sleep Quality total mean score | From enrollment to the end of the Mindfulness and Web-Based Physical Activity Program at 14 weeks
  Pittsburgh sleep quality index (PSQI) scores range from 0 to 21 points. A total score greater than 5 indicates "poor sleep quality".
Self-Confident Approach, Optimistic Approach, Helpless Approach, Submissive Approach, and Seeking of Social Support total mean score | From enrollment to the end of the Mindfulness and Web-Based Physical Activity Program at 14 weeks
  The 30-item Coping style scale (CSS) consists of a total of five subscales: Self-Confident Approach, Optimistic Approach, Helpless Approach, Submissive Approach, and Seeking of Social Support. The scale is evaluated based on its subdimensions. The scale has no total score. The total scores to be obtained from the sub-dimensions are as follows: 21 for self-confident approach, 15 for optimistic approach, 24 for helpless approach, 18 for submissive approach, and for 12 for seeking of social support. In the evaluation of the scale, the increase in scores obtained from the factors of self-confident, optimistic, and seeking of social support indicates that coping with stress is effective; whereas the increase in scores obtained from the factors of helpless approach and submissive approach shows that ineffective methods are being used to cope with stress. A high score on the sub-dimensions indicates that the individual uses the respective approach more frequently.

SECONDARY OUTCOMES:
Cardiovascular Risk | From enrollment to the end of the Mindfulness and Web-Based Physical Activity Program at 14 weeks
  This algorithm is used to calculate the 10-year cardiovascular disease risk of patients. As recommended in the QRISK*3 algorithm (https://www.qrisk.org/). If the QRISK3 score is > 20, it is classified as high risk; between 10-20%, it is classified as moderate risk; and <10 is classified as low risk.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Lok, Prof. Dr, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University Faculty of Medicine Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No